CLINICAL TRIAL: NCT02816879
Title: Improving Screening Tools to Better Predict High-Grade Anal Dysplasia for MSM
Brief Title: Anal Cytology Collection Procedures in Predicting High-Grade Anal Dysplasia in Men Who Have Sex With Men
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RCA169508A; NCI-2014-01292 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); JCCCID370 (Other: UCLA / Jonsson Comprehensive Cancer Center); RCA169508A (Other: UCLA / Jonsson Comprehensive Cancer Center); R01CA169508 (NIH); 13-000997 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2016-05-23; First posted 2016-06-29 (Estimated); Last update posted 2025-07-29 (Actual); Status verified 2024-07

CONDITIONS: Anal Carcinoma; HIV Infection; Human Papillomavirus Infection
MeSH Terms: conditions — Anus Neoplasms; HIV Infections; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Screening (anal cytology collection) (Experimental): Patients undergo anal cytology collection using 2 NF swabs and 1 Dacron swab for analysis via Pap staining, HPV genotyping, and PCR.
  Interventions: Procedure: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Cytology Specimen Collection Procedure — Undergo anal cytology collection
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This clinical trial compares three anal cytology collection procedures (collected at a single visit) in men who have sex with men (MSM). It also compares two different tests for human papilloma virus, the virus that causes high grade anal dysplasia, which is thought to occur before anal cancer. This study may help doctors develop better screening for high-grade anal dysplasia in MSM in order to identify those who need to return for additional screening and treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the sensitivity & specificity, predictive positive value (PPV), & predictive negative value (PNV) (test characteristics) & cellularity, beta-globin, deoxyribonucleic acid (DNA), ribonucleic acid (RNA), & protein (quality measures) from nylon-flocked (NF)- & Dacron-swab protocols to detect biopsy-detected high-grade anal intraepithelial neoplasia (HG-AIN) & human papillomavirus (HPV)-infections, using randomized-controlled study design.

II. Evaluate the test characteristics for anal cancer screening algorithms that incorporate sequentially or simultaneously performed high-threshold molecular HPV tests, with & without cytology, to predict HG-AIN.

III. Evaluate the cost-effectiveness & relative cost of single- & multiple-test anal cancer screening algorithms.

OUTLINE:

Patients undergo anal cytology collection using 2 NF swabs and 1 Dacron swab for analysis via Papanicolaou (Pap) staining, HPV genotyping, and polymerase chain reaction (PCR).

ELIGIBILITY:
Inclusion Criteria:

* Males who self-identify as having had or currently having sex with men; both human immunodeficiency virus (HIV)-infected and HIV-uninfected subjects are being enrolled

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of cytology specimens for Dacron swab compared to flocked nylon (NF) swab in predicting histology outcome | Baseline
  Two contingency tables will contrast cytology classification (for each swab type) with anal intraepithelial neoplasia (AIN) diagnosis based upon high-resolution anoscopy (HRA) & histology.

SECONDARY OUTCOMES:
Ability of APTIMA-HPV to predict risk for HG-AIN | Baseline
  Two contingency tables will contrast HPV infection characteristics for APTIMA-HPV & HC-2 compared to PCR based genotyping using Linear Array assay. Kappa statistics will be estimated to evaluate the observed versus expected agreement between the Linear Array assay (gold standard) & the findings for APTIMA-HPV & HC-2, separately. Prevalence estimates for 37 individual HPVs will be estimated from the data; also, for each type, agreement between the NF- & Dacron protocols for HPV genotypes will be summarized in tabular & graphical form.
Ability of Hybrid-capture 2 to predict risk for HG-AIN | Baseline
  Two contingency tables will contrast HPV infection characteristics for APTIMA-HPV & HC-2 compared to PCR based genotyping using Linear Array assay. Kappa statistics will be estimated to evaluate the observed versus expected agreement between the Linear Array assay (gold standard) & the findings for APTIMA-HPV & HC-2, separately. Prevalence estimates for 37 individual HPVs will be estimated from the data; also, for each type, agreement between the NF- & Dacron protocols for HPV genotypes will be summarized in tabular & graphical form.
Cost effectiveness analysis evaluating differences in survival, the cost of out-patient procedures & in-patient hospitalizations for invasive anal cancer. | Up to 3 years
  The cost-effectiveness analyses calculate incremental cost-effectiveness ratios (ICERs) comparing two intervention groups/strategies to the current standard of care, Dacron cytology alone. The ICER is the ratio of the difference in the total costs per patient between groups (numerator) versus the difference in quality-adjusted life-years (QALY) between groups (denominator). Specifically, for these analyses, ICERs are separately estimated for best single & best combination screening algorithm relative to usual care (Dacron-cytology). The analysis focuses on life-time costs.

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Wiley, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Los Angeles Gay and Lesbian Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Desert AIDS Project, Palm Springs, California